CLINICAL TRIAL: NCT00609050
Title: Self-Regulated Exercise in CF: A Randomized Trial
Brief Title: Exercise Training Study for Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, David Orenstein, Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR009285 (NIH); R01NR009285 (NIH)
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; exercise; perceived exertion; aerobic fitness; lung function; health related quality of life; self-regulated exercise
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Self-Regulated Exercise with Telephone Reinforcement
  Interventions: Behavioral: Self-Regulated Exercise with Telephone Reinforcement; Behavioral: Qualitative Approach
- 2 (Active Comparator): Attention Control
  Interventions: Behavioral: Standard Treatment; Behavioral: Qualitative Approach

INTERVENTIONS:
Behavioral: Self-Regulated Exercise with Telephone Reinforcement — The self-regulated exercise with telephone reinforcement group will engage in a three-times-a-week (or more) at home exercise regimen for 6 months during which they may choose the mode of exercise. They will receive weekly telephone calls about exercise and airway clearance. After 6 months, they will be instructed to maintain their self-regulated exercise activity for the remaining 6 months of the study, but they will not receive telephone calls
  Arms: 1
Behavioral: Standard Treatment — The attention control group will receive standard recommendations for exercise activity, during the first 6 months, as is common in our clinic. Also during the first 6 months, they will receive weekly telephone calls about airway clearance. For the final 6 months of the study, the attention control group will cross over to self-regulated exercise without telephone reinforcement.
  Arms: 2
Behavioral: Qualitative Approach — A qualitative naturalistic approach is nested within the primary experimental framework to explore the experiences of the children and parents, in both groups, with the exercise regimen.

SUMMARY:
The aim of this study is to test the effect of a 6-month program of self-regulated, home-based exercise with telephone reinforcement on the cardiorespiratory fitness, pulmonary function and health-related quality of life of children with cystic fibrosis (CF), compared to controls. Exploring the exercise experiences of the children and parents is a secondary aim.

DETAILED DESCRIPTION:
CF is a life-long illness that requires complex and dynamic adjustment by the patient and family. The nursing role is vital to the multidisciplinary team approach required in providing comprehensive, individualized care for these patients. Nurses facilitate the coordination of health care efforts and support the patient and family across physical and psychosocial domains. With the well-documented correlation between exercise tolerance and both survival and HRQoL, exercise represents a critical treatment focus for CF patients. Nurses contribute to standard exercise rehabilitation programs, through education, psychosocial support, and communication. In this exercise training study, the nursing role will include: a) teaching the patients and families how to use the OMNI scale, b) confirming that they understand the home-based exercise regimen, and c) ensuring that the home-care program is properly followed by placing weekly telephone calls to assess progress and barriers. Long-term nursing application will occur via dissemination of the OMNI training manual, to be developed as part of this study, for use by CF nurses in clinics worldwide.

ELIGIBILITY:
Inclusion Criteria:

* CF diagnosis
* age 10-18 years
* reliable pulmonary function tests
* living at home
* able to read
* able to ride a stationary bike
* able to walk and/or run on a treadmill.

Exclusion Criteria:

* Enrolled in another intervention study
* in structured aerobic activity for 30 continuous minutes 3 times per week
* sibling enrolled in study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Fitness: Peak VO2 | 1 year

SECONDARY OUTCOMES:
Cardiopulmonary fitness: VO2150 and peak power output | 1 year
Pulmonary function: FEV1 and sustained phonation time | 1 year
Health-related quality of life: Quality of well-being scale and cystic fibrosis questionnaire | 1 Year
Exercise experiences of children and parents: Interviews | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: David M Orenstein, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Antiono J & Janet Palumbo Cystic Fibrosis Center; Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided